CLINICAL TRIAL: NCT07140432
Title: Diagnostic Interest of Bone Tomoscintigraphy in the Search for Cervical Pseudarthrosis
Acronym: BOSCAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A00659-38
Record Dates: First submitted 2025-08-11; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cervical Pseudarthrosis
Keywords: cervical pseudarthrosis; imagining; hydric bone imagining; bone bridges; CT scans; diagnosis; cervical pain; bone scintigraphy; clinical presentation; diagnostic value
MeSH Terms: conditions — Disease; Neck Pain

STUDY DESIGN:
Masking Description: The scintigraphy examination will be interpreted, after reconstruction, on a via medical console (Siemens healthcare®) by two nuclear medicine physicians, blind to each other and to clinical data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scintigraphy (Experimental)
  Interventions: Other: Bone scintigraphy

INTERVENTIONS:
Other: Bone scintigraphy — A bone scintigraphy exam will be performed in addition of the already performed scanner in the current practice

SUMMARY:
Cervical pseudarthrosis is a classic complication and a challenge for challenge for spine surgeons. The rate of pseudarthrosis can range from 3 to 15%, and depend greatly on the patient, the approach the number of levels operated on.

Although some patients remain asymptomatic, most require revision surgery instability, cervical or radicular pain. Diagnosis of cervical pseudarthrosis remains difficult. The clinical presentation is non-specific, and there is no consensus on the imaging imaging. Radiographic evaluation lacks sensitivity. The dynamic images require prior calibration and anatomical landmarks difficult to visualize. Angle measurement lacks reproducibility and sensitivity. CT scans, currently considered the gold standard as the gold standard, provides valuable morphological data but does not provide information on the functional nature of bone bridges the functional nature of bone bridges and apparent consolidation, particularly incomplete.

At the same time, functional imaging using bone scintigraphy has been historically limited by lack of spatial resolution, absence of anatomical and radiation attenuation for deep structures.The advent of hybrid imaging makes it possible to these limitations. Recently, the 6 to 16 scanners fitted to gamma cameras enable a detailed study correlations between functional and anatomical data.

Interpretation criteria remain unestablished, however, and only one study reports the use of hydric bone imaging in the study of cervical pseudarthrosis. All patients were positive on scintigraphy. However, given the absence of "healthy" patients and the small number of patients the diagnostic value of bone scintigraphy in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 21 years of age
* Patients who have undergone cervical arthrodesis and are being treated at Clinique de la Sauvegarde or Clinique Convert
* Patients with a NDI clinical score at 1 year greater than 5
* Patient affiliated to/ or beneficiary of a Social Security scheme as definied by the law

Exclusion Criteria:

* Patients whose clinical condition requires rapid treatment that can't wait for examinations to be carried out
* Pregnancy and breastfeeding
* Protected person (curatorship, guardianship, safeguard of justice)
* History of hypersensitivity to the active substance ( sodium oxidronate) or to any of its constituents

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluating the sensitivity, specificity and positive predictive value of bone scintigraphy to diagnose cervical pseudarthrosis compared to the reference method | 12 months
  Sensitivity, specificity, and positive predictive value (PPV) will be evaluated against the reference method (based on intraoperative observation of hypermobility in cases of surgical revision and/or follow-up at 6 months (+/-1 month) and 12 months (+/-1 month) in the absence of surgical revision).

SECONDARY OUTCOMES:
Comparison of the sensitivity, specificity, and positive predictive value (PPV) of CT-scan versus bone scintigraphy in diagnosing cervical pseudarthrosis | 12 months
  Sensitivity, specificity, and positive predictive value (PPV) of CT-scan will be evaluated against the reference method (based on intraoperative observation of hypermobility in cases of surgical revision and/or follow-up at 6 months (+/-1 month) and 12 months (+/-1 month) in the absence of surgical revision) and then compared to the results for bone scintigraphy using a McNemar comparison as well as a Chi-2 test.
Assess the ability of scintigraphy to predict the probability of final consolidation in symptomatic patients at one year post arthrodesis | 12 months
  Final consolidation will be defined by the presence of bone bridges greater than 4 mm in at least two of the three sectors (anterior, middle, posterior) based on CT scan data at 2 years post-surgery.
  For the assessment of the probability of final consolidation, hyperfixation of at least one bone bridge greater than 4 mm wide (over its entire height), limited to one of the three sectors (anterior, middle, posterior) without the pseudarthrosis criteria described above, will be defined as a good probability of final consolidation. The presence of bone bridges more than 4 mm wide, over their entire height, with or without hyperfixation in at least two of the three sectors, will be defined as good consolidation

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Convert ( INA), Bourg-en-Bresse, France

IPD SHARING:
Plan to Share IPD: No